CLINICAL TRIAL: NCT00416988
Title: Skin Self-Examination for Early Detection of Melanoma: Intervention and Consequence
Brief Title: Educational Program in Skin Self-Examination To Detect Melanoma in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000454855; RIH-R01-CA78800
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2008-07

CONDITIONS: Melanoma (Skin); Weight Changes
Keywords: melanoma; weight changes
MeSH Terms: conditions — Melanoma; Body Weight Changes | interventions — Early Intervention, Educational

INTERVENTIONS:
Other: educational intervention

SUMMARY:
RATIONALE: An educational program may be effective in increasing monthly skin self-examinations to detect melanoma in healthy participants.

PURPOSE: This randomized clinical trial is studying how well an educational program works in increasing monthly skin self-examinations to detect melanoma in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of monthly thorough skin self-examinations (TSE) for early detection of melanoma in healthy participants who are under routine care by their primary care physician.
* Determine the impact of the intervention package and the resulting change in TSE performance, in terms of visits to healthcare providers for skin problems, in these participants.
* Evaluate the efficacy of this intervention package in improving performance of TSE in these participants.
* Estimate potential effect of this intervention on health care resource use.

OUTLINE: This is a controlled, randomized study.

Two weeks prior to their appointment with their physician, participants undergo a baseline assessment. During the appointment, participants are randomized to 1 of 2 intervention arms.

* Arm I (control): Participants receive written educational materials and watch a video on healthy dietary habits during their appointment. They receive nutrition tip sheets, including information related to reducing fat, saturated fat, and cholesterol in the diet, at 2 and 6 months after their initial appointment. Participants also undergo telephone assessments at 2, 6, and 12 months after their initial appointment.
* Arm II (skin self-examinations): Participants undergo a 10- to 15-minute face-to-face counseling session with the study intervention specialist and receive training in thorough skin self-examination (TSE) directly after their appointment. They also receive written educational materials and watch a 25-minute video designed to motivate and teach them to do TSE. Two weeks later, participants receive a follow-up call from the same study intervention specialist. Participants receive tailored feedback at 2 and 6 months and a motivational postcard at 4 months after their initial appointment. Participants also undergo telephone assessments as in arm I.

Participating physicians seeing participants in both arms attend a 60-minute educational session regarding skin cancer detection, prevention, identification, and triage, supplemented by written materials. They are also trained and prompted to deliver a 30-second message emphasizing the desirability of performing monthly TSE during their appointment with participants.

After completion of the study intervention, participants are offered the educational materials of the intervention arm to which they were not randomized.

PROJECTED ACCRUAL: A total of 1,135 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants who are scheduled for a routine or health maintenance visit with a participating primary care office that meets all of the following criteria:

  * At least 50% of patients are being seen for regular ongoing general medical care
  * Specializes in internal medicine (subspecialties allowed), family medicine, or obstetrics/gynecology
  * Employs at least 2 physicians who meet all of the following requirements:

    * Agree to participate
    * Work full-time, defined as at least 8 sessions per week of 3 or more hours
    * Completed post-graduate training
    * Not a federal employee or full-time hospital-based faculty
    * Have been in practice at least 1 year
    * Not planning on relocating or retiring within the next 3 years

PATIENT CHARACTERISTICS:

* Must be able to read in either English or Spanish
* Has no household member who has been previously enrolled on this study, including a person who has the same telephone number or address
* Not in acute discomfort
* Able to comply with intervention
* No impairment that would preclude skin self-examination
* Must be able to view video
* No illness or disability that would preclude participation in the study interview

PRIOR CONCURRENT THERAPY:

* Must not have been previously enrolled on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1135 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Weinstock, MD, PhD, Study Chair — Rhode Island Hospital

REFERENCES:
- [Result] Lee KB, Weinstock MA, Risica PM. Components of a successful intervention for monthly skin self-examination for early detection of melanoma: the "Check It Out" trial. J Am Acad Dermatol. 2008 Jun;58(6):1006-12. doi: 10.1016/j.jaad.2008.03.008. Epub 2008 Apr 11. PMID 18406492